CLINICAL TRIAL: NCT01411033
Title: Poznan Prospective Study of Type 1 Diabetic Patients Treated With Intensive Insulin Therapy From the Onset of the Disease.
Brief Title: Poznan Prospective Study of Type 1 Diabetic Patients
Acronym: PoProStu
Status: Active, not recruiting | Type: Observational
Sponsor: Poznan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Aleksandra Uruska, Prof. Dorota Zozulinska -Ziolkiewicz, Poznan University of Medical Sciences
Other Study IDs: 05/08/2003
Record Dates: First submitted 2011-08-02; First posted 2011-08-05 (Estimated); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Microangiopathy; Macroangiopathy; Insulin Treatment Overcorrection; Insulin Resistance
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Newly diagnosed diabetes mellitus type 1

SUMMARY:
The purpose of this study is to evaluate the development and progression of chronic complications (retinopathy, neuropathy, diabetic chronic renal disease, cardiovascular events) in patients with type 1 diabetes treated from the onset of the disease with recommended method of intensive insulin therapy. All patients attended a five-day structured training program during first hospitalization and re-education once year during the observation. After five years of observation and next - once a year chronic complications are assessed. The investigators would like to evaluate also the relationship of the management of the disease, knowledge about the treatment and diabetes, insulin resistance and inflammatory markers with development and progression of chronic complications.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed type 1 diabetes mellitus with features of complete insulin deficiency (serum C-peptide level <0.05 ng/ml, acetonuria, blood gases disturbances such as: pH <7.30, BE< -6 mmol/l, HCO3 <18 mmol/l)
* Age < 35 years old
* Educational course in intensive insulin therapy started at the onset of the disease after treatment of ketoacidosis
* Written consent

Exclusion Criteria:

* Uncertain type of diabetes mellitus
* Kidney failure (serum creatinine level > 1.1 mg/dl)
* Liver dysfunction (AspAt > 31 U/l, AlAt > 34 U/l)
* Acute inflammatory process
* Other concomitant diseases (i.e. neoplasm)

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: 100 Caucasian patients with newly diagnosed type 1 diabetes admitted to the Department of Internal Medicine and Diabetology, Poznan University of Medical Sciences in years 1994-1999, treated from the onset of the disease with intensive insulintherapy.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 1994-01; Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Retinopathy | 1 year
Diabetic chronic renal disease | 1 year
Neuropathy | 1 year
Cardiovascular events | 1 year
  stroke, heart infarct, death

SECONDARY OUTCOMES:
Metabolic management of diabetes | 1 year
  HbA1c, hypoglycaemic episodes, lipid profile, blood pressure, BMI
Quality of life | 1 year
Intima media thickness | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Dorota A Zozulinska-Ziolkiewicz, Prof, Principal Investigator — Department of Internal Medicine and Diabetology, Poznan University of Medical Sciences

REFERENCES:
- [Result] Wegner M, Piorunska-Stolzmann M, Araszkiewicz A, Zozulinska-Ziolkiewicz D, Naskret D, Uruska A, Wierusz-Wysocka B. Does oxidized LDL contribute to atherosclerotic plaque formation and microvascular complications in patients with type 1 diabetes? Clin Biochem. 2012 Dec;45(18):1620-3. doi: 10.1016/j.clinbiochem.2012.08.019. Epub 2012 Aug 29. PMID 22960236
- [Result] Wegner M, Piorunska-Stolzmann M, Araszkiewicz A, Zozulinska-Ziolkiewicz D, Wierusz-Wysocka B. Evaluation of paraoxonase 1 arylesterase activity and lipid peroxide levels in patients with type 1 diabetes. Pol Arch Med Wewn. 2011 Dec;121(12):448-54. PMID 22157813
- [Result] Araszkiewicz A, Uruska A, Zozulinska-Ziolkiewicz D, Pilacinski S, Wierusz-Wysocka B. Factors related to insulin resistance in type 1 diabetic patients treated with intensive insulin therapy from the onset of the disease. Diabetes Res Clin Pract. 2010 Nov;90(2):e23-4. doi: 10.1016/j.diabres.2010.05.010. Epub 2010 Jun 11. No abstract available. PMID 20541277
- [Result] Wegner M, Araszkiewicz A, Zozulinska-Ziolkiewicz D, Wierusz-Wysocka B, Piorunska-Mikolajczak A, Piorunska-Stolzmann M. The relationship between concentrations of magnesium and oxidized low density lipoprotein and the activity of platelet activating factor acetylhydrolase in the serum of patients with type 1 diabetes. Magnes Res. 2010 Jun;23(2):97-104. doi: 10.1684/mrh.2010.0207. Epub 2010 May 27. PMID 20507838
- [Result] Uruska A, Araszkiewicz A, Zozulinska-Ziolkiewicz D, Uruski P, Wierusz-Wysocka B. Insulin resistance is associated with microangiopathy in type 1 diabetic patients treated with intensive insulin therapy from the onset of disease. Exp Clin Endocrinol Diabetes. 2010 Aug;118(8):478-84. doi: 10.1055/s-0030-1249635. Epub 2010 Apr 6. PMID 20373280
- [Result] Wegner M, Araszkiewicz A, Piorunska-Mikolajczak A, Zozulinska-Ziolkiewicz D, Wierusz-Wysocka B, Piorunska-Stolzmann M. The evaluation of IL-12 concentration, PAF-AH, and PLA(2) activity in patients with type 1 diabetes treated with intensive insulin therapy. Clin Biochem. 2009 Nov;42(16-17):1621-7. doi: 10.1016/j.clinbiochem.2009.07.023. Epub 2009 Aug 3. PMID 19651120
- [Result] Araszkiewicz A, Zozulinska-Ziolkiewicz D, Trepinska M, Wierusz-Wysocka B. Knowledge after five-day teaching program in intensive insulin therapy performed at the onset of type 1 diabetes influence the development of late diabetic complications. Diabetes Res Clin Pract. 2008 Jul;81(1):61-7. doi: 10.1016/j.diabres.2008.02.009. Epub 2008 Apr 2. PMID 18378034
- [Result] Araszkiewicz A, Zozulinska D, Trepinska M, Wierusz-Wysocka B. [Is intensive functional insulin therapy the method of choice in newly diagnosed type-1 diabetes mellitus?]. Pol Merkur Lekarski. 2004 Nov;17(101):463-6. Polish. PMID 15754632
- [Result] Uruska A, Araszkiewicz A, Zozulinska-Ziolkiewicz D, Wegner M, Grzelka A, Wierusz-Wysocka B. Does serum cystatin C level reflect insulin resistance in patients with type 1 diabetes? Clin Biochem. 2014 Sep;47(13-14):1235-8. doi: 10.1016/j.clinbiochem.2014.06.014. Epub 2014 Jun 20. PMID 24956263
- [Result] Uruska A, Araszkiewicz A, Uruski P, Zozulinska-Ziolkiewicz D. Higher risk of microvascular complications in smokers with type 1 diabetes despite intensive insulin therapy. Microvasc Res. 2014 Mar;92:79-84. doi: 10.1016/j.mvr.2014.01.002. Epub 2014 Jan 12. PMID 24423616
- [Result] Grzelka A, Naskret D, Araszkiewicz A, Uruska A, Wegner M, Zozulinska-Ziolkiewicz D. Higher concentrations of osteoprotegerin in type 1 diabetic patients are related to retinopathy: Results from the Poznan Prospective Study. Adv Clin Exp Med. 2017 Dec;26(9):1343-1349. doi: 10.17219/acem/65072. PMID 29442454
- [Result] Uruska A, Niedzwiecki P, Araszkiewicz A, Zozulinska-Ziolkiewicz D. Brain-derived neurotrophic factor and insulin resistance during hyperinsulinaemic-euglycaemic clamp in type 1 diabetes patients in the PoProStu. Diabetes Metab. 2017 Oct;43(5):472-474. doi: 10.1016/j.diabet.2016.12.007. Epub 2017 Jan 27. No abstract available. PMID 28139435
- [Result] Grzelka A, Araszkiewicz A, Uruska A, Zozulinska-Ziolkiewicz D. Prevalence of anti-thyroid peroxidase in adults with type 1 diabetes participating in Poznan Prospective Study. Adv Clin Exp Med. 2015 Jan-Feb;24(1):79-84. doi: 10.17219/acem/38149. PMID 25923090
- [Result] Araszkiewicz A, Naskret D, Zozulinska-Ziolkiewicz D, Pilacinski S, Uruska A, Grzelka A, Wegner M, Wierusz-Wysocka B. Skin autofluorescence is associated with carotid intima-media thickness, diabetic microangiopathy, and long-lasting metabolic control in type 1 diabetic patients. Results from Poznan Prospective Study. Microvasc Res. 2015 Mar;98:62-7. doi: 10.1016/j.mvr.2015.01.002. Epub 2015 Jan 10. PMID 25582078
- [Result] Araszkiewicz A, Zozulinska-Ziolkiewicz D, Pilacinski S, Naskret D, Uruska A, Wierusz-Wysocka B. Baseline diabetic knowledge after 5-day teaching program is an independent predictor of subclinical macroangiopathy in patients with type 1 diabetes (Poznan Prospective Study). Adv Med Sci. 2014 Sep;59(2):240-4. doi: 10.1016/j.advms.2013.12.005. Epub 2014 Jun 9. PMID 25090481